CLINICAL TRIAL: NCT07031349
Title: Evaluation of Changes in Upper Airway Dimensions and Subjective Sleep Quality Following Miniscrew-Assisted Rapid Palatal Expansion: A Questionnaire-Based Study
Brief Title: MARPE-Associated Changes in Sleep and Airway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Responsible Party: Principal Investigator, Seda Sağoğlu, Research Assistant, Konya Necmettin Erbakan Üniversitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025/596
Record Dates: First submitted 2025-06-11; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rapid Maxillary Expansion
Keywords: MARPE; STOP-BANG; PSQI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MARPE (Other): Adult individuals treated with miniscrew-assisted rapid palatal expansion (MARPE)
  Interventions: Device: MARPE

INTERVENTIONS:
Device: MARPE — Adult patients with maxillary constriction underwent maxillary expansion using a miniscrew-assisted rapid palatal expander (MARPE).

SUMMARY:
At the beginning of MARPE treatment (T1) and at the end of the 3-month consolidation phase (T2), patients will complete the teen-STOP-BANG questionnaire and the Pittsburgh Sleep Quality Index (PSQI) to assess the potential benefit of MARPE in reducing the risk of obstructive sleep apnea syndrome (OSAS).

Additionally, changes in the upper airway will be evaluated using CBCT images obtained at T1 and T2.

DETAILED DESCRIPTION:
In this clinical routine, approximately 30% of patients requiring rapid maxillary expansion (RME) are treated using the MARPE (Miniscrew-Assisted Rapid Palatal Expansion) method. To evaluate the potential benefits of MARPE in reducing the risk of obstructive sleep apnea syndrome (OSAS), patients are asked to complete the teen-STOP-BANG questionnaire and the Pittsburgh Sleep Quality Index (PSQI) at the beginning of treatment (T1) and at the end of the 3-month consolidation phase (T2).

To determine whether patients should undergo MARPE or conventional RME, midpalatal suture maturation is assessed as part of the routine protocol using cone-beam computed tomography (CBCT) images obtained before treatment initiation (T1). At the end of the MARPE screw activation period, a follow-up CBCT scan is routinely obtained to evaluate potential complications such as fractures in the zygomatic buttress region, alveolar bending, and the presence of dehiscence or fenestration on root surfaces. This scan also facilitates the controlled initiation of prolonged fixed orthodontic treatment.

Additionally, CBCT images obtained at T1 and T2 will be used to measure and compare the dimensions of the upper airway, including both oropharyngeal and nasopharyngeal regions.

ELIGIBILITY:
Inclusion Criteria:

Class I malocclusion Maxillary transverse deficiency Age between 15 and 18 years No systemic disease, cleft lip and palate, or speech disorders No history of prior orthodontic treatment Voluntary agreement to participate in the study Good oral hygiene ANB angle between 2° and 5°

Exclusion Criteria:

Presence of systemic diseases Smoking Poor oral hygiene Lack of cooperation Mental retardation Obesity or nutritional disorders Macroglossia or mandibular retrognathia

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-05 (Estimated)

PRIMARY OUTCOMES:
Change in obstructive sleep apnea (OSA) risk as measured by the teen-STOP-BANG questionnaire | 3 month
  The teen-STOP-BANG questionnaire will be used to assess changes in OSA risk following MARPE treatment. STOP-BANG scores range from 0 to 8; a score of at least 3 indicates that the patient is at risk of OSAHS, and a score of at least 5 indicates that the patient is at high risk of OSA.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of surgically assisted rapid maxillary expansion on obstructive sleep apnea. — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=Effect+of+surgically+assisted+rapid+maxillary+expansion+on+obstructive+sleep+apnea&btnG=